CLINICAL TRIAL: NCT00306787
Title: A Multicenter, Randomized, Double-blind Study to Compare the Efficacy and Safety of Patient-initiated Famciclovir 1000 mg b.i.d. x 1 Day to Valacyclovir 500 mg b.i.d. x 3 Days in Immunocompetent Adults With Recurrent Genital Herpes
Brief Title: Efficacy and Safety of Famciclovir 1-day Treatment Compared to 3-day Treatment With Valacyclovir in Adults With Recurrent Genital Herpes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFAM810A2308
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Genital Herpes
Keywords: Herpes simplex; genital herpes; famciclovir; valacyclovir; Recurrent genital herpes
MeSH Terms: conditions — Herpes Genitalis; Herpes Simplex | interventions — Famciclovir; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Famciclovir (Experimental): Patients received Famciclovir 1000 mg (2 x 500 mg tablets) twice a day for one day. The first dose was to be taken within 6 hours after onset of prodromal symptoms or genital herpes lesions and the second dose approximately 12 hours later. Patients also received 1 valacyclovir placebo capsule, beginning with the first famciclovir dose, twice a day for 3 days, each taken about 12 hours apart.
  Interventions: Drug: Famciclovir; Drug: Placebo matching valacyclovir
- Valacyclovir (Active Comparator): Patients received Valacyclovir 500 mg capsule twice a day approximately 12 hours apart for 3 consecutive days. The first dose was to be taken within 6 hours after onset of prodromal symptoms or genital herpes lesions. On the first day patients also received 2 famciclovir placebo tablets taken with the first 2 doses of Valacyclovir.
  Interventions: Drug: Valacyclovir; Drug: Placebo matching famciclovir

INTERVENTIONS:
Drug: Famciclovir — Famciclovir 500 mg tablet
  Other Names: Famvir
  Arms: Famciclovir
Drug: Valacyclovir — Valacyclovir 500 mg capsule
  Other Names: Valtrex
  Arms: Valacyclovir
Drug: Placebo matching famciclovir — Famciclovir placebo, matching in size, color and forms of famciclovir tablet.
  Arms: Valacyclovir
Drug: Placebo matching valacyclovir — Valacyclovir placebo, matching in size, color and forms of valacyclovir capsule.
  Arms: Famciclovir

SUMMARY:
This study will assess the safety and efficacy of one-day famciclovir (1000 mg twice a day (b.i.d)) in reducing the duration of genital herpes lesions and the associated symptoms compared to three-day treatment with valacyclovir (500 mg capsule b.i.d).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* History of at least 4 recurrences of genital herpes in the preceding 12 months
* Lesions located on the external genitalia or anogenital region
* Willing to discontinue suppressive treatment
* Documented positive herpes simplex virus (HSV)
* General good health, and history of normal renal function

Exclusion Criteria:

* Women of childbearing potential not using approved form of contraceptive
* Pregnant or nursing women
* History of hypersensitivity to famciclovir, valacyclovir, or acyclovir
* Known to be immunosuppressed
* Known to have renal dysfunction
* Receiving anti-herpes therapy
* Known to have other genital tract disorders
* Known to have condition which could interfere with drug absorption

Additional protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1179 (Actual)
Dates: Start 2006-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (65):
- United States (51):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Novartis Investigative Site, Chandler, Arizona
  - Women's Health Research, Phoenix, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - NEA Women's Clinic, Jonesboro, Arkansas
  - The Woman's Clinic, Little Rock, Arkansas
  - Providence Clinical Research, Burbank, California
  - Dermatology Research Associates, Los Angeles, California
  - Sacramento Research Medical Group, Sacramento, California
  - North California Research Corp., Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Conant Research, San Francisco, California
  - Barbara Davis Center, Denver, Colorado
  - Cohen & Womack, P.C., Lakewood, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - International Research Association LLC, Miami, Florida
  - Orlando Clinical Research Ctr., Orlando, Florida
  - Avancia Research, Pembroke Pines, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Medisphere Medical Research Center, LLC., Evansville, Indiana
  - Indiana University Infectious Disease Research Group, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Common Wealth Biomedical Research, Madisonville, Kentucky
  - SNBL Clinical Pharmacology Center, Baltimore, Maryland
  - Future Care Studies, Springfield, Massachusetts
  - Clayton Research Institute, St Louis, Missouri
  - Deaconess Billings Clinic Research Center, Billings, Montana
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - UNC Clinical Research., Raleigh, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Providence Health Partners-Center for Clinical Research, Dayton, Ohio
  - Lynne Health Science Institute, Oklahoma City, Oklahoma
  - Westover Heights Clinic, Portland, Oregon
  - Paddington Testing Co. Inc, Philadelphia, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - S. Carolina Clinical Research Center, Columbia, South Carolina
  - Research Inc., Florence, South Carolina
  - Palmetto Clinical Trial Services, LLC, Simpsonville, South Carolina
  - Benchmark Research, Austin, Texas
  - Renaissance Clinical Research and Hypertension Clinic, Dallas, Texas
  - Center for Clinical Studies (TX Medical Center), Houston, Texas
  - Center for Clinical Studies, Houston, Texas
  - University of Utah-School of Medicine (Div. of Inf. Disease), Salt Lake City, Utah
  - Salt Lake Women's Center/Physician's Research Options, Sandy City, Utah
  - Clinical Trials of Virginia, Inc., Richmond, Virginia
  - University of Washington, Virology Research Clinic, Seattle, Washington
  - Liberty Research Center, Tacoma, Washington
- Novartis Investigative Site, Darlinghurst, New South Wales, Australia
- Canada (8):
  - Novartis Investigational Site, Edmonton, Alberta
  - Novartis Investigational Site, Vancouver, British Columbia
  - Novartis Investigational Site, Winnipeg, Manitoba
  - Novartis Investigational Site, Markham, Ontario
  - Novartis Investigational Site, Ottawa, Ontario
  - Novartis Investigational Site, Laval, Quebec
  - Novartis Investigational Site, Montreal, Quebec
  - Novartis Investigational Site, Sainte-Foy, Quebec
- Germany (5):
  - Novartis Investigational Site, Augsburg
  - Novartis Investigational Site, Berlin
  - Novartis Investigational Site, Freiburg im Breisgau
  - Novartis Investigational Site, Rostock
  - Novartis Investigational Site, Wolfsburg

REFERENCES:
- [Derived] Bodsworth N, Fife K, Koltun W, Tyring S, Abudalu M, Prichard M, Hamed K. Single-day famciclovir for the treatment of genital herpes: follow-up results of time to next recurrence and assessment of antiviral resistance. Curr Med Res Opin. 2009 Feb;25(2):483-7. doi: 10.1185/03007990802664678. PMID 19192993
- See also: eRecruitment — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=520

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1179 patients were randomized in the study and followed to their first genital herpes recurrence. A total of 423 patients did not experience a recurrence within 4 months of randomization therefore, no treatment was initiated and study drug was not taken. A total of 756 patients were randomized and took study drug (safety population).
Groups:
- Valacyclovir: Patients received Valacyclovir 500 mg capsule twice a day (b.i.d) approximately 12 hours apart for 3 consecutive days. The first dose was to be taken within 6 hours after onset of prodromal symptoms or genital herpes lesions. On the first day patients also received 2 famciclovir placebo tablets taken with the first 2 doses of Valacyclovir.
Period: Overall Study
Arm/Group | Famciclovir | Valacyclovir
Started | 579 | 600
Received Study Drug (Safety Population) | 371 | 385
Intent to Treat (ITT) Population | 370 | 381
Completed | 345 | 359
Not Completed | 234 | 241
Not completed — Discontinued without taking study drug | 208 | 215
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 8 | 10
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Lost to Follow-up | 9 | 6
Not completed — Administrative problems | 4 | 0
Not completed — Abnormal laboratory value(s) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Famciclovir | Valacyclovir | Total
Number analyzed (Participants) | 370 | 381 | 751
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data is provided for the intent to treat (IIT) population, which included all randomized patients who initiated treatment with (i.e. received any dose of) the study drug, with the intention of treating genital herpes recurrences.
  years | 39.6 (11.6) | 41.7 (12.6) | 40.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 243 | 488
  Male | 125 | 138 | 263

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Time to Healing of All Non-aborted Genital Herpes Lesions
Description: Time to healing of all non-aborted genital herpes lesions was defined as the time from the first dose of study drug taken no earlier than the recurrence of genital herpes to the investigator-assessed time of healing (i.e. loss of all crusts and re-epithelialization of the lesions; erythema could have been present). Non-aborted lesions are lesions which underwent vesicle, ulcer/soft crust, and/or hard crust formation and required re-epithelialization for healing. The median time was estimated using Kaplan-Meier method by censoring missing values at the time of last clinical lesion observation.
Time Frame: 72 hours after initiation of study medication up to Day 20
Population: Modified Intent To Treat (mITT) population. The mITT population included all patients who initiated treatment with the study drug, with the intention of treating genital herpes recurrences who developed non-aborted genital herpes lesions during the treated recurrence except those with confirmed aborted lesions at the final clinical assessment.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Famciclovir | Valacyclovir
Number analyzed (Participants) | 249 | 253
days | 4.25 [3.06 to 5.78] | 4.08 [3.02 to 5.80]
Statistical Analysis 1: Comparison: Famciclovir vs Valacyclovir; Difference in time to healing= time to healing for famciclovir- time to healing for valacyclovir; Test type: Non-Inferiority or Equivalence — The estimated power for non-inferiority test (90%) was based on the non-inferiority margin of 1.0 day; Hodges-Lehman; Median Difference (Final Values) = 0.16, 95% CI 2-sided [-0.15 to 0.60]

2. Secondary Outcome: Percentage of Participants With Aborted Genital Herpes Lesions
Description: Lesions that developed no further than the papule stage (erythema may have been present) were considered as aborted lesions. Prodrome also was considered the sign of aborted lesions in this study. Lesions which underwent vesicle, ulcer/soft crust, and/or hard crust formation and required re-epithelialization for healing were considered as non-aborted lesions.
Time Frame: 72 hours after initiation of study medication up to Day 20
Population: ITT population. Patients who discontinued from the study before healing of non-aborted lesions was confirmed and patients who completed the study after 21 days since treatment initiation without non-aborted lesion stages and without a final assessment on aborted lesion status were assumed to have non-aborted lesions in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Famciclovir | Valacyclovir
Number analyzed (Participants) | 370 | 381
Percentage of participants
  Aborted Lesions | 32.7 | 33.6
  Non-Aborted lesions | 67.3 | 66.4

3. Secondary Outcome: Investigator-assessed Time to Healing of All (Non-aborted and Aborted) Genital Herpes Lesions
Description: Lesions that developed no further than the papule stage (erythema may have been present) were considered as aborted lesions. Prodrome also was considered the sign of aborted lesions in this study. Lesions which underwent vesicle, ulcer/soft crust, and/or hard crust formation and required re-epithelialization for healing were considered as non-aborted lesions. The median time was estimated using Kaplan-Meier method.
Time Frame: 72 hours after initiation of study medication up to Day 20
Population: ITT population. Median time was estimated by kaplan-Meier method by censoring the missing non-aborted times at last clinical observation. Patients with aborted lesions were assigned a time to healing of zero.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Famciclovir | Valacyclovir
Number analyzed (Participants) | 370 | 381
days | 3.07 [0.00 to 5.00] | 3.01 [0.00 to 4.88]

4. Secondary Outcome: Time to Resolution of Symptoms Associated With Recurrent Genital Herpes
Description: Kaplan-Meier estimated time in hours of the resolution of all symptoms (pain, burning, itching, tingling and tenderness) associated with recurrent genital herpes. Kaplan-Meier method is used to estimate the time to resolution of symptoms.
Time Frame: 72 hours after initiation of study medication up to Day 20
Population: ITT population. If the resolution of any or all symptoms was not confirmed by a subsequent visit or diary entry, the time to resolution was censored at the time of the last diary entry. If a patient dropped out before any diary entries were created, the patient was assigned a censoring time of 0. n= number of patients with symptoms.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Famciclovir | Valacyclovir
Number analyzed (Participants) | 370 | 381
hours
  Pain (n = 220, 228) | 18.0 [0.0 to 52.7] | 20.3 [0.00 to 46.6]
  Burning (n = 221, 218) | 16.1 [0.0 to 50.5] | 12.6 [0.0 to 47.5]
  Itching (n = 309, 297) | 43.9 [12.2 to 76.7] | 43.5 [11.5 to 85.6]
  Tingling (n = 266, 275) | 23.8 [0.0 to 58.0] | 23.0 [0.0 to 50.5]
  Tenderness (n = 298, 311) | 55.2 [20.4 to 106.0] | 48.0 [14.3 to 87.3]

5. Secondary Outcome: Number of Patients With a Second Recurrence of Genital Herpes
Description: Patients who experienced a first recurrence of genital herpes and took study medication were followed for a period of up to 6 months to the second recurrence.
Time Frame: Up to 6 months after investigator assessed healing of first recurrence of genital herpes
Population: ITT population included all randomized patients who initiated treatment with (i.e. received any dose of) the study drug, with the intention of treating genital herpes recurrences.
Measure: Number; unit: participants
Arm/Group | Famciclovir | Valacyclovir
Number analyzed (Participants) | 370 | 381
participants
  Patients continued in follow up period | 324 | 342
  Patients with 2nd recurrence in follow up period | 226 | 231

6. Secondary Outcome: Time to a Second Recurrence of Genital Herpes
Description: Patients who experienced a first recurrence of genital herpes and took study medication were followed for a period of up to 6 months to the second recurrence. Time to a second recurrence of genital herpes was calculated in 2 ways as follows:
  1. From the date of treatment initiation no earlier than the recurrence of genital herpes to the date of onset for the second recurrence, or
  2. From the date of healing of non-aborted lesions or confirmation of aborted lesions to the date of onset for the second recurrence.
Time Frame: Up to 6 months after investigator assessed healing of first recurrence of genital herpes
Population: ITT population. Patients with missing time-to-second recurrence were not included in the calculation of the median.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Famciclovir | Valacyclovir
Number analyzed (Participants) | 226 | 231
days
  From treatment initiation | 33.5 [18 to 67] | 38.0 [18 to 73]
  From date of healing /confirmation | 27.5 [14 to 63] | 32.0 [14 to 69]

ADVERSE EVENTS:
Time Frame: 30 days post last dose of study medication
Description: Safety Population
Arm/Group | Famciclovir | Valacyclovir
Serious Adverse Events (participants affected / at risk) | 2/371 | 1/385
Other Adverse Events (participants affected / at risk) | 66/371 | 47/385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Famciclovir (N=371) | Valacyclovir (N=385)
Myocardial ischemia (Cardiac disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0
Substance Abuse (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Famciclovir (N=371) | Valacyclovir (N=385)
Headache (Nervous system disorders) | 29 | 17
Nausea (Gastrointestinal disorders) | 23 | 18
Diarrhea (Gastrointestinal disorders) | 8 | 5
Vomiting (Gastrointestinal disorders) | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.